CLINICAL TRIAL: NCT07197827
Title: A Phase 1/2, Multicenter, Open-Label, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of YL242 Monotherapy and Combinations in Advanced Solid Tumors.
Brief Title: A Study of YL242 in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YL242-INT-101-01
Record Dates: First submitted 2025-09-26; First posted 2025-09-29 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor
Keywords: Oncology; VEGF; Antibody drug conjugate; Developmental Phase I/II
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 and Part 2: Mono Dose Escalation & Expansion (Experimental): Participants receive YL242 administered via intravenous (IV) solution per protocol defined dose level and frequency.
  Interventions: Drug: YL242
- Part 3 and 4: Combination Dose Escalation & Expansion (Experimental): Participants receive YL242 at protocol defined dose level, in combination with Pembrolizumab (200 mg), administered via intravenous (IV) solution at protocol defined dose level and frequency.
  Interventions: Drug: YL242; Pembrolizumab
- Part 5: Combination Dose Optimization and Expansion (Experimental): Participants receive YL242, 5-FU and LV, administered via intravenous (IV) solution.
  Interventions: Drug: YL242; 5-FU; LV
- Part 6: Combination Dose Optimization and Expansion (Experimental): Participants receive YL242, pembrolizumab and 5-FU, administered via intravenous (IV) solution at protocol defined frequency.
  Interventions: Drug: YL242; Pembrolizumab; 5-FU

INTERVENTIONS:
Drug: YL242 — The YL242 drug product is provided as a lyophilized powder containing 200 mg of YL242 in a glass vial. The initial dose of YL242 will be infused IV into each patient for 90±10 minutes. If there is no infusion-related reaction after the initial dose, the second and subsequent doses of YL242 will be infused IV into each patient for 60±10 minutes.
  Arms: Part 1 and Part 2: Mono Dose Escalation & Expansion
Drug: YL242; Pembrolizumab — The YL242 drug product is provided as a lyophilized powder containing 200 mg of YL242 in a glass vial. The initial dose of YL242 will be infused IV into each patient for 90±10 minutes. If there is no infusion-related reaction after the initial dose, the second and subsequent doses of YL242 will be infused IV into each patient for 60±10 minutes. Pembrolizumab will be administered subsequent to YL242.
  Arms: Part 3 and 4: Combination Dose Escalation & Expansion
Drug: YL242; 5-FU; LV — The YL242 drug product is provided as a lyophilized powder containing 200 mg of YL242 in a glass vial. The initial dose of YL242 will be infused IV into each patient for 90±10 minutes. If there is no infusion-related reaction after the initial dose, the second and subsequent doses of YL242 will be infused IV into each patient for 60±10 minutes.
  LV and 5-FU will be sequentially administered following YL242.
  Arms: Part 5: Combination Dose Optimization and Expansion
Drug: YL242; Pembrolizumab; 5-FU — The YL242 drug product is provided as a lyophilized powder containing 200 mg of YL242 in a glass vial. YL242 will be administered via Intravenous (IV) Infusion.
  Pembrolizumab and 5-FU will be administered in sequence after YL242.
  Arms: Part 6: Combination Dose Optimization and Expansion

SUMMARY:
This is a multicenter, open-label study to evaluate the safety and tolerability of YL242 monotherapy and combination in participants with advanced solid malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1
* Adequate organ and bone marrow function
* Tumor type:

Part 1-3: Advanced/unresectable or metastatic solid malignant tumor; Have received at least one prior line of systemic anti-tumor therapy

Part 4: locally advanced or metastatic non-sq NSCLC without AGA and HCC; Have not received any systemic anti-tumor therapy;

Part 5: mCRC, have received at least one (5a) or one (5b) prior line of systemic anti-tumor therapy

Part 6: advanced or metastatic HER2-negative G/GEJ; have received at least one (6a) or one (6b) prior line of systemic anti-tumor therapy

Exclusion Criteria:

* Be intolerant to prior treatment with a topoisomerase I inhibitor or an ADC that consists of a topoisomerase I inhibitor
* Uncontrolled or clinically significant cardiovascular and cerebrovascular diseases
* Clinically significant concomitant pulmonary disease
* A history of leptomeningeal carcinomatosis or carcinomatous meningitis
* Any illness, medical condition, organ system dysfunction, or social situation, including but not limited to mental illness or substance/alcohol abuse, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, adversely affect the patient's ability to cooperate and participate in the study, or compromise the interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) in Participants With Advanced Solid Malignant Tumors (Part 2, and 4-6) | Approximately within 36 months
  Objective response rate (ORR) was defined as the proportion of participants who achieve either complete response [CR] or partial response [PR] per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Number of Participants Reporting Treatment-emergent Adverse Events (TEAEs) | Baseline up to 42 days post last patients last dose, approximately within 36 months
  AEs will be collected systematically from signing of the informed consent form (ICF) through 42 days after last dose.

SECONDARY OUTCOMES:
Area Under the Serum Concentration Time Curve (AUC) of YL242 | Approximately within 36 months
Maximum Plasma Concentration (Cmax) of YL242 | Approximately within 36 months
Time to Maximum Plasma Concentration (Tmax) of YL242 | Approximately within 36 months
Incidence of anti-YL242 antibody | Approximately within 36 months
Terminal Elimination Half-life (t1/2) of Serum YL242 | Approximately within 36 months
Disease Control Rate (DCR) | Approximately within 36 months
  Disease control rate (DCR) was calculated as the proportion of participants demonstrating complete response (CR), partial response (PR), or stable disease.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (7):
  - US-201, New Haven, Connecticut
  - US-202, Sarasota, Florida
  - US-204, Boston, Massachusetts
  - US-206, Grand Rapids, Michigan
  - US-205, Nashville, Tennessee
  - US-203, Houston, Texas
  - US-207, San Antonio, Texas
- Australia (5):
  - AUS-101, Liverpool, New South Wales
  - AUS-102, Darlinghurst, Victoria
  - AUS-104, Fitzroy, Victoria
  - AUS-103, Heidelberg, Victoria
  - AUS-105, Nedlands, Western Australia
- China (3):
  - CN-303, Harbin, Heilongjiang
  - CN-301, Shanghai, Shanghai Municipality
  - CN-302, Hangzhou, Zhejiang